CLINICAL TRIAL: NCT02160236
Title: Comparison of Postoperative Analgesic Efficacy of Intravenous Dexketoprofen Trometamol With Tenoxicam in Lumbar Disc Surgery
Brief Title: Comparison of Postoperative Analgesic Efficacy of Intravenous Dexketoprofen Trometamol With Tenoxicam
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Nazife Küçük, resident, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2013/469
Record Dates: First submitted 2014-06-08; First posted 2014-06-10 (Estimated); Last update posted 2014-11-10 (Estimated); Status verified 2014-11

CONDITIONS: Postoperative Pain
Keywords: dexketoprofen trometamol; tenoxicam; postoperative pain
MeSH Terms: conditions — Pain, Postoperative | interventions — dexketoprofen trometamol; tenoxicam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- dexketoprofen trometamol (Active Comparator): before end of the surgery via intravenous administration 50 mg dexketoprofen trometamol in 0.9 % NaCl 100 cc
  Interventions: Drug: dexketoprofen trometamol
- tenoxicam (Active Comparator): before the end of the surgery via administration intravenous 20 mg tenoxicam in 0.9% NaCl in 100 cc
  Interventions: Drug: tenoxicam
- serum physiologic (Placebo Comparator): before end of the surgery via administration intravenous 0.9 % NaCl 100 cc
  Interventions: Drug: serum physiologic

INTERVENTIONS:
Drug: dexketoprofen trometamol — before end of the surgery via intravenous administration 50 mg dexketoprofen trometamol in 0.9 % NaCl 100 cc
  Other Names: arveles
  Arms: dexketoprofen trometamol
Drug: tenoxicam — before the end of the surgery via administration intravenous 20 mg tenoxicam in 0.9% NaCl in 100 cc
  Other Names: oksamen
  Arms: tenoxicam
Drug: serum physiologic — before end of the surgery via administration intravenous 0.9 % NaCl 100 cc
  Arms: serum physiologic

SUMMARY:
In this study the investigators aimed to compare of postoperative analgesic effects of intravenous dexketoprofen trometamol and tenoxicam in lumbar disc surgery.

DETAILED DESCRIPTION:
Lumbar disc surgery is associated with moderate to severe back and radicular pain postoperatively which has unfavorable effects on patients recovery and procedures outcome. Dexketoprofen has been reported to be one of the NSAİDs that can provide good results when compared with narcotics in many painful conditions and especially in the treatment of the moderate to severe postoperative pain that may develop after lumbal disc surgery. Tenoxicam is a thienothiazine derivative of the oxicam class of NSAİDs. There are some studies in which NSAİDs have been used to together with opioids for postoperative analgesia showing that they decrease opioid consumption and side effects

ELIGIBILITY:
Inclusion Criteria:

* ASA 1-2
* between 18-65 age
* elective lumbar disc surgery

Exclusion Criteria:

* history of gastrointestinal bleeding
* peptic ulcer disease
* bleeding disorders
* history of allergic reactions to NSAİDs
* chronic pain syndrome

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2014-11; Primary Completion 2015-02 (Estimated); Study Completion 2015-02 (Estimated)

PRIMARY OUTCOMES:
analgesic consumption | postoperative 1 day
  morphine consumption (patient control analgesia procedure) was recorded

SECONDARY OUTCOMES:
visual analog scale | postoperative 1 day
  visual analog scale on rest and movement was recorded

CONTACTS AND LOCATIONS:
Overall Officials: nazife küçük, resident, Principal Investigator — TC Erciyes University
Locations (1):
- Erciyes Universty Hospital, Kayseri, Turkey (Türkiye)